CLINICAL TRIAL: NCT02463370
Title: Effectiveness of Four Versus Ten Local Anesthetic Injections for Post-submucosal Resection Pain Relief: a Randomized, Double Blinded Clinical Trial
Brief Title: Four vs. Ten Local Anesthetic Injections for SMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 122014
Record Dates: First submitted 2015-05-13; First posted 2015-06-04 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Submucosal Resection of the Nasal Septum (SMR)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group II (Experimental): Group II patients will receive local anesthetic infiltration in two injections on each side of the face at the maxillary and infra-orbital areas and the remaining injections are placebo (saline).
  Interventions: Other: suprazygomatic maxillary area infiltration; Other: non-suprazygomatic maxillary area placebo
- Group V (Experimental): Group V patients will receive local anesthesia in five injections on each side of the face at the infra-orbital area, supratrochlear area, medial to the medial canthus, nasal still and anterior septum. The remaining maxillary injection is placebo.
  Interventions: Other: non-suprazygomatic maxillary area infiltration; Other: suprazygomatic maxillary area placebo

INTERVENTIONS:
Other: suprazygomatic maxillary area infiltration — Local anesthetic infiltration in two injections on each side of the face at the maxillary and infra-orbital areas.
  Arms: Group II
Other: non-suprazygomatic maxillary area placebo — The remaining injections at supratrochlear area, medial to the medial canthus, nasal still and anterior septum are placebo (saline)
  Arms: Group II
Other: non-suprazygomatic maxillary area infiltration — Local anesthetic infiltration in five injections on each side of the face at the infra-orbital area, supratrochlear area, medial to the medial canthus, nasal still and anterior septum.
  Arms: Group V
Other: suprazygomatic maxillary area placebo — The remaining maxillary injection is placebo.
  Arms: Group V

SUMMARY:
Submucosal resection of the nasal septum (SMR) could be performed under local anesthetic infiltration performed through ten injections in addition to general anesthesia which was associated with less postoperative pain and shorter hospital stay.

However, the local infiltration technique is time-consuming and requires a large number of facial injections. This gave rise to the idea of reducing the number of injections while retaining the effectiveness of the local anesthetic technique.

Decreasing the number of injections could be achieved by blocking the superior maxillary nerve (V2) and the infra-orbital nerve since it would result in anesthetizing the surgical area as well after induction of general anesthesia.

The purpose of this prospective double-blind clinical trial was to compare the effectiveness of four versus ten local anesthetic injections in terms of postoperative pain relief. The secondary objective was to compare patients' and surgeons' satisfaction between the two techniques.

DETAILED DESCRIPTION:
Informed consent will be obtained from patients (ASA I and II) scheduled to undergo elective submucosal resection of the nasal septum between May and November 2015.

The sealed envelope technique is used to randomly assign patients into two groups. The anesthetists, surgeons, and nurses who collected the will be blinded to the study groups. Patients in both groups will receive general anesthesia and six injections on each side of the face at the following points: suprazygomatic maxillary (V2) area, infra-orbital area, supratrochlear area, medial to the medial canthus, nasal still and anterior septum. Group II patients will receive local anesthetic infiltration in two injections on each side of the face at the maxillary and infra-orbital areas and the remaining injections are placebo (saline). Group V patients will receive local anesthesia in five injections on each side of the face at the infra-orbital area, supratrochlear area, medial to the medial canthus, nasal still and anterior septum. The remaining maxillary injection is placebo.

To maintain double-blindness, three syringes (one 5 ml and two 10 ml) will be used for the six injections. They are prepared by a nurse who is not involved in the study. The 5 ml syringe (Becton Dickinson, Franklin Lakes New Jersey, USA) is labeled "F" indicating that it should be used at the infra-orbital area for both groups. The total injected solution is about 2 ml. One of the 10 ml syringes (Becton Dickinson, Franklin Lakes New Jersey, USA) is labeled "I" indicating that it should be used for infiltration at the supratrochlear area, medial to the medial canthus, nasal still and anterior septum. The total injected solution is 6 ml. The second 10 ml syringe is labeled "Z" to be used for the suprazygomatic maxillary nerve block.

The syringe labeled "F" always contains the local anesthetic solution. When syringe "I" contains the anesthetic mixture (group V), then syringe "Z" is placebo. In contrary, when syringe "Z" contains the anesthetic solution (group II), syringe "I" is placebo. The local anesthetic mixture is composed of 3 ml lidocaine 2%, 3 ml bupivacaine 0.5%, and 1 ml fentanyl 50 µg/ml. In addition, syringe "F" contains 50 µg clonidine while syringes "I" and "Z" have 100 µg clonidine (when they contain the anesthetic solution).

* Suprazygomatic maxillary nerve block technique:

The needle is inserted perpendicular to the skin and advanced to reach the greater wing of the sphenoid. The needle is then angulated at 200 and 100 in the anterior and caudal directions respectively. The needle is advanced about 3-3.5 cm through the pterygopalatine fossa. The total amount of injected solution is 0.1 ml/kg with a maximum volume of 3.5 ml on each side of the face.

* General anesthesia technique:

Induction of general anesthesia is achieved by using 1-2 mg/kg propofol, 1-1.5 µg/kg intravenous fentanyl and 2-3 ml midazolam. Endotracheal intubation is facilitated by 0.5 mg/kg atracurium. Anesthesia is maintained using 1-1.5% sevoflurane, 0.5-0.75 µg/kg/hr fentanyl, 70% nitrous oxide and 30% oxygen. Any hemodynamic change of ±25% from pre-induction values results in a gradual increase or decrease of the sevoflurane concentration.

* Surgical procedure:

Following preparation and draping of the nose, the septum is infiltrated using a solution of xylocaine with 1% adrenaline. This would facilitate vasoconstriction and hydrodissection. A hemitransfixion incision is made in which the mucoperiosteal and mucoperichondrial flaps are elevated and then the deviated septum is resected. The flaps are sutured (Vicryl sutures) and packed with two Merocel packs. The patients will be asked to visit the clinic after 48 hours to remove the packs.

* Data collection:

Data will be collected at predetermined time intervals by trained nurses. Patients will be followed-up for ten postoperative days and contacted daily through phone calls after hospital charge.

Mean arterial pressure (MAP) and heart rate (HR) are collected preoperatively, before incision and post incision. Monitoring devices are pulse oximeter and noninvasive arterial blood pressure. Postoperative pain is assessed at rest using the Numeric Rating Scale. The number of patients who will consume analgesics is recorded. Pain scores, incidence of oozing, headache, edema, hematoma, toothache, as well as postoperative nausea and vomiting (PONV) are collected during the first postoperative day every six hours (at 0, 6 and 12 hours) and after that once daily for the next nine days. Postoperative oozing is defined as changing three nasal dressings in 24 hours.

Patients' and surgeons' satisfaction will be asked to rate their satisfaction on a four point scale (very satisfied, satisfied, little satisfied or dissatisfied). Surgeon satisfaction is based on intraoperative hemodynamic stability of the patient and bleeding. Postoperative surgeon satisfaction is dependent on patients' feeling of pain (especially upon pack removal), bleeding and number of phone calls made to the surgeon. Surgeons are asked to generally recall the number of calls.

Patients' satisfaction is based on their postoperative comfort determined by their feeling of pain, headache and PONV.

* Postoperative pain management:

During the first 6 hours only, 1-1.5 mg/kg intravenous tramadol hydrochloride is given if the pain score was four or greater. If the score was less than four, patients are given 1 g intravenous perfalgan. After the first six postoperative hours, patients are given two tablets 500 mg oral paracetamol if the pain score is less than four. In case paracetamol is not sufficient, patients are prescribed 100 mg Voltarene, a non-steroidal anti-inflammatory drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients 15 years and older

Exclusion Criteria:

* Patients younger than 15 years old or have the following: a history of allergy to local anesthetics, suspected malignant neoplasm, BMI>40 kg/m2, hemodynamic instability or infection at the site of injection.
* Patients whom it will not be possible to follow them through telephone calls will also be excluded.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain over ten days measured by the Numeric Rating Scale | First postoperative day every six hours (at 0, 6 and 12 hours) and after that once daily for the next nine days
  Numeric Rating Scale will be used to measure postoperative pain

SECONDARY OUTCOMES:
Patients' satisfaction | Patients' satisfaction at 0, 6 and 12 hours postoperatively.
  Patients' satisfaction is based on their postoperative comfort determined by their feeling of pain, headache and PONV. It will be measured using four point scale (very satisfied, satisfied, little satisfied or dissatisfied)
Surgeons' satisfaction | Surgeons' satisfaction intraoperatively and postoperatively
  Surgeon satisfaction is based on intraoperative hemodynamic stability of the patient and bleeding. Postoperative surgeon satisfaction is dependent on patients' feeling of pain (especially upon pack removal), bleeding and number of phone calls made to the surgeon. It will be assessed using four point scale (very satisfied, satisfied, little satisfied or dissatisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon